CLINICAL TRIAL: NCT03974789
Title: Discriminant Capacity and Thresholds of Salivary Cortisol in Chemiluminescence in the Diagnosis of Hypercorticisms: Phase III Diagnostic Evaluation Study
Brief Title: Discriminant Capacity and Thresholds of Salivary Cortisol in Chemiluminescence in the Diagnosis of Hypercorticisms
Acronym: COSHING
Status: Active, not recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: NIMAO/2018-03/DPDB-01
Record Dates: First submitted 2019-06-03; First posted 2019-06-05 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Cushing Disease
MeSH Terms: conditions — Pituitary ACTH Hypersecretion | interventions — Hematologic Tests; Urinalysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Suspected Cushing Disease
  Interventions: Diagnostic Test: Blood test; Diagnostic Test: 24-hour Urine test; Diagnostic Test: Saliva swab; Diagnostic Test: Dexamethasone test

INTERVENTIONS:
Diagnostic Test: Blood test — Plasma cortisol level test
Diagnostic Test: 24-hour Urine test — Urinary free cortisol test
Diagnostic Test: Saliva swab — salivette® for salivary cortisol quantification
Diagnostic Test: Dexamethasone test — Dectancyl® 2 x 0.5 mg tablets (total 1 mg)

SUMMARY:
Automated immunodosage methods (Roche Elecsys cortisol and IDS cortisol dosing kits) offer a simple and inexpensive technology routinely used in a medical biology laboratory. They can be used to define robust diagnostic thresholds for salivary cortisol for the diagnosis of Cushing's syndrome and pseudo-Cushing combining the three tests performed as part of the patient's usual management. (ie two urinary free cortisol (UFC), the dexamethasone suppression test, and Diurnal variation of plasma cortisol).

ELIGIBILITY:
Inclusion Criteria:

* The patient is under consultation in the department of metabolic and endocrine disorders at the CHU Nimes for diagnosis or follow-up of hypercortisol assessment
* The patient must be a member or beneficiary of a health insurance plan

Exclusion Criteria:

* The patient is pregnant, parturient or breastfeeding
* The patient has a cardiovascular or metabolic state against the indication of dexamethasone

  - Patient with DFG < 30 ml/min/1.73 m2
* The patient has suffered urinary incontinence rendering 24-hour urinary collection impossible or non-interpretable
* The patient has a urinary catheter
* The patient is taking corticoids (oral, inhaled, intra-venous or cutaneous)

  .Patient exposed to interfering treatments (Itraconazole, ritonavir, megestrol acetate, medroxyprogesterone acetate, TSH, estrogen-progestogen pill, hormonal coil)
* The subject is in a period of exclusion determined by a previous study
* The subject opposes their participation in the study
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The target population of the study is patients suspected of hypercorticism. The study's source population will correspond to all patients (men and women) between the ages of 18 and 65 hospitalized in the metabolic and endocrine disorders department of CHU Nîmes for hypercorticism assessment in primary diagnosis or in a follow-up report.
Sampling Method: Non-Probability Sample
Enrollment: 380 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Salivary cortisol measured by Roche Elecsys cortisol kit | Day 1 (at screening)
  nmol/l
Salivary cortisol measured by IDS cortisol dosing kit at screening | Day 1 (at screening)
  nmol/l

SECONDARY OUTCOMES:
Salivary cortisol measured by Roche Elecsys cortisol kit | Day 2 and Day 3
  nmol/l
Salivary cortisol measured by IDS cortisol dosing kit | Day 2 and Day 3
  nmol/l
Salivary cortisol measured measured by LC-MS/MS | Day 1, 2 and 3
  nmol/l
Dexamethasone suppression test | Day 4
  µg/l and nmol/l (cut-off for diagnosis: 50nmol/l)
Diurnal variation of plasma cortisol | Day 3
  Roche Elecsys cortisol kiet; µg/l and nmol/l (cut-off for diagnosis: 200nmol/l)
Urinary free cortisol | Day 3
  Radioimmunoassay; µg/l and nmol/l

CONTACTS AND LOCATIONS:
Overall Officials: David de Brauwere, Principal Investigator — CHU Nimes
Locations (1):
- CHU de Nimes, Nîmes, France